CLINICAL TRIAL: NCT01145846
Title: A Prospective Randomized Comparison of Idarubicin and High-dose Daunorubicin in Combination With Cytarabine in the Induction Chemotherapy for Acute Myeloid Leukemia
Brief Title: Idarubicin Versus High Dose Daunorubicin in Acute Myelogenous Leukemia (AML)
Acronym: AIvsAD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cooperative Study Group A for Hematology (Network)
Responsible Party: COSAH, Cooperative Study Group A for Hematology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C-022
Record Dates: First submitted 2010-05-19; First posted 2010-06-17 (Estimated); Last update posted 2010-06-17 (Estimated); Status verified 2010-06

CONDITIONS: Acute Myelogenous Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine; Daunorubicin; Idarubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (AI regimen) (Experimental): Cytarabine 200 mg/m2/day by continuous iv infusion over 24 hours daily for 7 days (D 1-7) plus Idarubicin 12 mg/m2/day iv daily for 3 days (D 1-3)
  Interventions: Drug: Cytarabine plus Daunorubicin [Arm II (AD regimen)]

INTERVENTIONS:
Drug: Cytarabine plus Daunorubicin [Arm II (AD regimen)] — Cytarabine 200 mg/m2/day by continuous iv infusion over 24 hours daily for 7 days (D 1-7) plus Daunorubicin 90 mg/m2/day iv daily for 3 days (D 1-3)
  Other Names: Cytarabine /Idarubicin

SUMMARY:
The purpose of this non-inferiority study is to compare the effectiveness of two induction chemotherapy regimens (cytarabine plus idarubicin [AI] versus cytarabine plus high-dose daunorubicin [AD]) in AML. The effectiveness will be evaluated in terms of complete remission (CR) rate.

DETAILED DESCRIPTION:
1. INDUCTION CHEMOTHERAPY

   * For patients randomized to receive Idarubicin (Arm I, AI regimen) will be given Cytarabine 200 mg/m2/day by continuous iv infusion over 24 hours daily for 7 days (D 1-7) along with Idarubicin 12 mg/m2/day iv daily for 3 days (D 1-3).
   * For patients randomized to receive Daunorubicin (Arm II, AD regimen) will be given Cytarabine 200 mg/m2/day by continuous iv infusion over 24 hours daily for 7 days (D 1-7) along with Daunorubicin 90 mg/m2/day iv daily for 3 days (D 1-3).
2. INTERIM BONE MARROW EXAMINATION

   * Bone marrow aspiration and biopsy will be done between 14 to 21 days after start of induction chemotherapy.
   * If the bone marrow is hypoplastic and contains no more than 5% blast cells, further chemotherapy will be deferred and the marrow examination will be repeated at the time of neutrophils over 1,000/mcL and platelets over 100,000/mcL in the peripheral blood for the evaluation of complete remission.
   * If more than 5% blast cells persist at interim or later repeated bone marrow examination, a course of re-induction chemotherapy will be given.
3. RE-INDUCTION CHEMOTHERAPY

   -Reinduction chemotherapy
   * Arm I (AI regimen) : Cytarabine 200 mg/m2/day by continuous iv infusion over 24 hours daily for 5 days (D 1-5) plus idarubicin 8 mg/m2/day iv daily for 2 days (D 1-2)
   * Arm II (AD regimen) : Cytarabine 200 mg/m2/day by continuous iv infusion over 24 hours daily for 5 days (D 1-5) plus Daunorubicin 45 mg/m2/day iv daily for 2 days (D 1-2) .Reinduction chemotherapy should be delayed if there is a significant infection or other co-morbid medical condition.
   * Patients who do not have a complete remission after a second course of induction chemotherapy will be removed from the study
4. POSTREMISSION CHEMOTHERAPY .The same postremission therapy will be given to the patients in both arms. .For patients with good- or intermediate-risk cytogenetic features or unknown cytogenetics (see appendix II), 4 courses of high-dose cytarabine will be given as post-remission therapy. Cytarabine 3 g/m2 will be administered in a 3-hour iv infusion every 12 hours on days 1, 3, and 5 (a total of six doses per course).

   .For patients with high-risk cytogenetic features (see appendix II), 4 courses of intermediate-dose Cytarabine plus Etoposide will be given as post-remission therapy. Cytarabine 1 g/m2 will be given in a 1-hour iv infusion on days 1 to 6 (a total of six doses per course) and Etoposide 150 mg/m2/day will be administered in a 5-hour iv infusion on days 1 to 3 (a total of three doses per course).

   .Sequential courses of postremission therapy will be given no sooner than every 28 days or 1 week after adequate marrow recovery.

   .Postremission chemotherapy should be delayed if there is a significant infection or other co-morbid medical condition.

   .One or two doses of Cytarabine can be omitted according to the attending physician's decision for the followings: .Marrow recovery requires more than 28 days.
   * A confluent maculopapular eruption or drug-induced desquamation
   * Photophobia or conjunctivitis unrelieved within 24 hours by ophthalmic steroid drops
   * More than 4 episodes of watery diarrhea per day
   * A fourfold increase in a previously normal serum aminotransferase or alkaline phosphatase level or a total bilirubin level exceeding 3.0 mg/dL .Treatment with high-dose cytarabine will be discontinued in patients with severe cerebellar ataxia, confusion, or other central nervous system signs thought to be unrelated to antiemetic medication.
5. EVALUATION DURING TREATMENT .During induction and consolidation chemotherapy: CBC with differentials (daily), chemical battery with electrolyte (twice a week), coagulation battery (once a week), chest x-ray (once a week).

   .Bone marrow examination will be repeated on day 15 of induction chemotherapy (for the evaluation of hypocellular marrow) and at the time of ANC ≥ 1,000/μl and platelets ≥ 100,000/μl in the peripheral blood (for the evaluation of complete remission). Chromosomal analysis will be repeated at the time of the evaluation of complete remission.
6. POST-TREATMENT FOLLOW-UP

   .After the completion of postremission treatment (i.e. following consolidation chemotherapy or HCT): CBC with differentials (monthly for the first 12 months, then every 2-3 months for the next 4 years), other studies such as MRD monitoring (as indicated)
7. TREATMENT EVALUATION *FFICACY EVALUATION

   * Complete remission (CR): Bone marrow blasts < 5%; absence of blasts with Auer rods; absence of extramedullary disease; absolute neutrophil count > 1,000/mcL; platelet count > 100,000/mcL; independence of red cell transfusion (Döhner H et al, 2010).
   * All criteria need to be fulfilled; marrow evaluation should be based on a count of 200 nucleated cells in an aspirate with spicules; if ambiguous, consider repeat exam after 5 to 7 days; flow cytometric evaluation may help to distinguish between persistent leukemia and regenerating normal marrow; a marrow biopsy should be performed in cases of dry tap, or if no spicules are obtained; no minimum duration of response required.
   * CR with incomplete recovery (CRi): All CR criteria except for residual neutropenia (< 1,000/mcL) or thrombocytopenia (< 100,000/mcL).
   * Cause of treatment failure
   * Resistant disease (RD): Failure to achieve CR or CRi; only includes patients surviving ≥ 7 days following completion of initial treatment, with evidence of persistent leukemia by blood and/or bone marrow examination.
   * Death in aplasia: Deaths occurring ≥ 7 days following completion of initial treatment while cytopenic; with an aplastic or hypoplastic bone marrow obtained within 7 days of death, without evidence of persistent leukemia.
   * Death from indeterminate cause: Deaths occurring before completion of therapy, or < 7 days following its completion; or deaths occurring ≥ 7 days following completion of initial therapy with no blasts in the blood, but no bone marrow examination available.
   * Relapse: Bone marrow blasts ≥ 5%; or reappearance of blasts in the blood; or development of extramedullary disease.
   * In cases with low blast percentages (5-10%), a repeat marrow should be performed to confirm relapse. Appearance of new dysplastic changes should be closely monitored for emerging relapse. In a patient who has been recently treated, dysplasia or a transient increase in blasts may reflect a chemotherapy effect and recovery of hematopoiesis. Cytogenetics should be tested to distinguish true relapse from therapy-related MDS/AML.

ELIGIBILITY:
Inclusion Criteria:

* Patients with previously-untreated acute myeloid leukemia (20% or more of blasts in bone marrow and/or blood; M6 subtype may have less than 20% of blasts.). Therapy-related leukemia or leukemia after myelodysplastic syndrome will be included.
* 15 years old or older, but 65 years or younger
* Adequate performance status (Karnofsky score of 50 or more)
* Adequate hepatic and renal function (AST, ALT, bilirubin and creatinine < 2.5 x upper normal limit). Elevation of AST or ALT due to hepatic infiltration of leukemic cells will be permitted.
* Adequate cardiac function (left ventricular ejection fraction of 45% or more on heart scan or echocardiogram)
* Signed and dated informed consent must be obtained

Exclusion Criteria:

* Patients with acute promyelocytic leukemia or bcr-abl gene rearrangement
* Patients with CNS leukemia
* Patients with primary granulocytic sarcoma without bone marrow involvement
* Prior chemotherapy for leukemia or anthracycline treatment for any malignancy. Hydroxyurea for reduction of leukemic cell burden before induction chemotherapy will be permitted.
* Presence of significant active infection
* Presence of uncontrolled bleeding
* Significant cardiovascular disease including myocardial infarction within previous 6 months
* Any coexisting major illness or organ failure
* Patients with psychiatric disorder or mental deficiency severe as to make compliance with the treatment unlike, and making informed consent impossible
* Nursing women, pregnant women, women of childbearing potential who do not want adequate contraception
* Patients with a diagnosis of prior malignancy unless disease-free for at least 5 years following therapy with curative intent (except curatively treated nonmelanoma skin cancer, in situ carcinoma, or cervical intraepithelial neoplasia)

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 316 (Estimated)
Dates: Start 2010-05; Primary Completion 2012-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Complete remission rate | five years
  A complete remission will be defined as blasts of 5% or less in a normocellular bone marrow with neutrophils of 1,000/mcL or more and platelets of 100,000/mcL or more in the peripheral blood, the disappearance of all blasts in the peripheral blood, and no evidence of extramedullary leukemic cell infiltration

SECONDARY OUTCOMES:
Duration of CR, relapse-free survival(RFS),event-free survival(EFS),Overall survival(OS) | Five years
  * This study will evaluate the impacts of induction chemotherapy regimen on duration of CR, relapse-free survival (RFS), event-free survival (EFS), and overall survival (OS).
  * This study will also evaluate the clinical significance of genetic polymorphisms of drug-metabolizing enzymes and mutations of leukemia-related genes.

CONTACTS AND LOCATIONS:
Overall Officials: Je Hwan Lee, Professor, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Songpa-gu, South Korea

REFERENCES:
- See also: A prospective randomized comparison of idarubicin and high-dose daunorubicin in combination with cytarabine in the induction chemotherapy for acute myeloid leukemia — http://www.google.co.kr